CLINICAL TRIAL: NCT05357417
Title: Utidelone Plus Bevacizumab for Advanced Breast Cancer With Brain Metastases: A Multicenter, Single Arm, Open Label, Phase II Trial
Brief Title: Utidelone Plus Bevacizumab for Advanced Breast Cancer With Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-MBC08-BM02
Record Dates: First submitted 2022-04-21; First posted 2022-05-02 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: brain metastases;bevacizumab;utidelone
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cohort 1 (Experimental): HER2-negative advanced breast cancer with brain metastases who have received at least one prior anthracycline and one prior taxane
  Interventions: Drug: utidelone; Drug: Bevacizumab
- cohort 2 (Experimental): HER2-positive advanced breast cancer with brain metastases who have failed trastuzumab and pyrotinib
  Interventions: Drug: utidelone; Drug: Bevacizumab

INTERVENTIONS:
Drug: utidelone — 30mg/m2 (±10%), day 1-5 every 3-week cycle
Drug: Bevacizumab — 15mg/kg, day 1

SUMMARY:
This study aims to investigate the efficacy and safety of utidelone in combination with bevacizumab in the treatment of advanced breast cancer with brain metastases, and thus provides a new systemic treatment strategy for those patients.

DETAILED DESCRIPTION:
This is a multicenter,open label, phase 2 trial to investigate the efficacy and safety of utidelone in combination with bevacizumab in the treatment of advanced breast cancer with brain metastases. Patients with HER2-negative advanced breast cancer who have received at least one prior anthracycline and one prior taxane or HER2-positive advanced breast cancer who have failed trastuzumab and pyrotinib, and with at least one measurable CNS lesion are eligible for the study.

This study includes 2 cohorts, and the Simon two-stage design are applied, respectively. A total of 48 patients with HER2-negative advanced breast cancer are included in cohort 1, and 52 patients with HER-2 positive patients are enrolled in cohort 2. Patients in both cohorts receive bevacizumab, 15mg/kg, day 1, and utidelone, 30mg/m2 (±10%), day 1-5 every 3-week cycle until disease progression or unmanageable toxicity. The primary endpoint is CNS-ORR according to the RECIST 1.1. The secondary endpoints include CNS-ORR according to RANO criteria, CNS-PFS assessed by investigator, extracranial ORR, extracranial PFS, OS, time to WBRT, quality of life and safety profile according to NCI-CTCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years; histologically or cytologically confirmed invasive breast cancer with metastatic disease; patients without pathologically or cytologically confirmed metastatic disease must have physical or radiological proof of metastasis;
2. With measurable CNS disease, defined as at least one parenchymal brain lesion that can be accurately measured in at least one dimension by local radiology;
3. Previously treated with at least one anthracycline and one taxane (as neoadjuvant therapy, adjuvant therapy, palliative therapy, or both);
4. Patients in cohort 2 have failed trastuzumab and pyrotinib treatment;
5. Prior unproven treatment progression with utidelone or bevacizumab;
6. ECOG PS of 0-1 and life expectancy exceeding 12 weeks;
7. Normal organ and bone marrow function; normal blood sample within one week before enrollment (as determined by the laboratory's normal values in each center), including WBC ≥ 3.0 x 109/L, ANC ≥ 1.5×109/L, PLT ≥ 100×109/L; normal kidney and liver function within one week before enrollment (as determined by the laboratory's normal values in each center), including TBIL ≤ 1.5 ULN, SGPT/ALT ≤ 2.5 ULN (≤ 5 ULN in patients with liver metastases), SGOT/AST ≤ 2.5 ULN, Ccr ≥ 60 ml/min;
8. Neurological lesions must be < grade 2 according to NCI CTCAE version 5.0 within four weeks before enrollment;
9. Without major organ dysfunction or heart disease;
10. Those of childbearing potential should use appropriate contraception before and during study period.

Exclusion Criteria:

1. Patients with leptomeningeal metastases who are not adequately treated by dehydration, hormone therapy, or urgently need radiotherapy;
2. Presence of effusions that cannot be controlled by drainage or other treatment (e.g., massive pericardial, thoracic, or abdominal effusions);
3. Patients received WBRT, chemotherapy, major surgery, targeted therapy or immunotherapy within two weeks before enrollment, received endocrine therapy within one week before enrollment, or received nitrosourea or mitomycin based chemotherapy within six weeks before enrollment；
4. Participation in another clinical trial within four weeks before enrollment；
5. History of grade 3 or 4 allergic events to bevacizumab or utidelone;
6. Contraindications to MRI gadolinium-based contrast agents, such as pacemakers, shrapnel or intraocular foreign bodies;
7. Other malignancies within three years, except for cured cervical carcinoma in situ, cutaneous basal cell carcinoma, or cutaneous squamous cell carcinoma;
8. More than two seizures within four weeks before enrollment;
9. Insufficiently controlled hypertension, or history of hypertensive crisis or hypertensive encephalopathy;
10. CNS hemorrhage of grade 2 or higher within 12 months before enrollment;
11. NYHA class II or severe congestive heart failure, or history of myocardial infarction or unstable angina within six months;
12. History of hemoptysis within six months before enrollment, or evidence of bleeding tendency or significant coagulation dysfunction within one month;
13. Receiving full dose of warfarin or equivalent currently, or using aspirin (325 mg/day) within ten days;
14. Needs for major surgery, open biopsy or with major trauma within 28 days or during the study period;
15. History of abdominal fistula or gastrointestinal perforation within six months；
16. Presence of unhealed wound, active ulcer or untreated fracture;
17. Any other condition inappropriate for this study deemed by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
CNS-ORR according to the RECIST 1.1. | up to 2 years
  the proportion of patients with the best intracranial response of confirmed complete or partial response according to RECIST 1·1, as assessed by the investigator

SECONDARY OUTCOMES:
CNS-ORR according to RANO criteria | up to 2 years
  the proportion of patients with the best intracranial response of confirmed complete or partial response according to RANO criteria, as assessed by the investigator
CNS-PFS assessed by investigator | up to 2 years
  time from the first dose to disease progression or any-cause death
extracranial ORR | up to 2 years
  proportion of patients with confirmed extracranial complete or partial response per RECIST 1·1
extracranial PFS | up to 2 years
  time from the first dose to disease progression or any-cause death
OS | Estimated up to 3 year
  time from the first dose of study drug to any-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification are available following article publication.
Supporting Information: Study Protocol
Time Frame: Three years from publication
Access Criteria: Please contact Central contact person by Email

REFERENCES:
- [Derived] Yan M, Lv H, Liu X, Wang S, Geng C, Song Y, Liu Z, Niu L, Zhang M, Wang C, Feng Y, Zeng H, Sun H, Wang J, Xiang Y, Tang L, Qiu R. Utidelone Plus Bevacizumab for ERBB2-Negative Metastatic Breast Cancer and Active Brain Metastases: The U-BOMB Phase 2 Nonrandomized Clinical Trial. JAMA Oncol. 2025 Aug 1;11(8):883-889. doi: 10.1001/jamaoncol.2025.1694. PMID 40569584